CLINICAL TRIAL: NCT04859608
Title: Personalized Spacing of Eculizumab Infusions Based on Therapeutic Pharmacological Monitoring: Prospective Health-economic Evaluation in Patients in Remission With Atypical Hemolytic Uraemic Syndrome Requiring Long-term Treatment.
Brief Title: Personalized Spacing of Eculizumab Infusions Based on Therapeutic Pharmacological Monitoring (EspacECU)
Acronym: EspacECU
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Tours (Other)
Collaborators: Centre Hospitalier Universitaire, Amiens (Other); University Hospital, Angers (Other Government); Centre Hospitalier Universitaire de Besancon (Other); University Hospital, Caen (Other); Centre Hospitalier of Chartres (Other); Nantes University Hospital (Other); University of Nancy (Other); Poitiers University Hospital (Other); Rennes University Hospital (Other); University Hospital, Rouen (Other); University Hospital, Strasbourg, France (Other); Centre Hospitalier Universitaire de Nice (Other); Hôpital Necker-Enfants Malades (Other); Tenon Hospital, Paris (Other); University Hospital, Lille (Other); Reims University hospital (Other); University Hospital, Clermont-Ferrand (Other); Assistance Publique Hopitaux De Marseille (Other); Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DR200088-EspacECU
Record Dates: First submitted 2021-02-02; First posted 2021-04-26 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Hemolytic-Uremic Syndrome, Atypical
Keywords: Hemolytic-Uremic Syndrome; Kidney Diseases; Thrombotic Microangiopathies; Therapeutic drug monitoring; Eculizumab tailoring; Cost-utility analysis; Markov model
MeSH Terms: conditions — Atypical Hemolytic Uremic Syndrome; Hemolytic-Uremic Syndrome; Kidney Diseases; Thrombotic Microangiopathies

STUDY DESIGN:
Intervention Model Description: Randomized (2:1) controlled study, open-label, with Markov modeling.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Therapeutic drug monitoring (Experimental): Tailored dosing schedule for eculizumab based on therapeutic drug monitoring
  Interventions: Drug: Spacing of Eculizumab infusions
- Control (No Intervention): Initial eculizumab schedule is continued (real-life arm). No eculizumab dosages are performed in this arm.

INTERVENTIONS:
Drug: Spacing of Eculizumab infusions — Personalized spacing of eculizumab infusions using a pharmacokinetic population model to estimate eculizumab concentration ( a one-week spacing of eculizumab infusion will be decide if predicted eculizumab concentration in the event of spacing is > 150 mg/L). Spacing of infusion can be decided every 3 months.
  Arms: Therapeutic drug monitoring

SUMMARY:
Eculizumab is an anti-C5 monoclonal antibody approved for rare diseases including atypical haemolytic-uraemic syndrome. The maintenance phase dosing regimen is identical for all adult patients but several studies have shown a high interindividual kinetics variability. A tailored administration of eculizumab based on therapeutic drug monitoring will be compared with real-life administration in adults suffering from an atypical haemolytic uraemic syndrome. The objective is to improve efficiency of eculizumab administration.

DETAILED DESCRIPTION:
Eculizumab is a very expensive drug (450 000 euros per year per patient). According to the usual administration scheme, the eculizumab is administrated by intravenous infusion, every 14 or 21 days in hospital. Studies have shown the possibility of extending the administration intervals in patients with a high concentration of eculizumab.

A personalized spacing of eculizumab infusions, based on a therapeutic drug monitoring, is expected to improve the patient's quality of life and lead to substantial savings.

For these reasons, the objective of this study is to explore the efficiency of a personalized spacing of eculizumab infusions compared to the usual administration scheme (without personalization) from the French health Insurance perspective. The efficiency will be assessed by estimating the incremental cost per QALY (Quality-Adjusted Life Year) gained at 18 months (duration of follow-up in the clinical trial) and at 5 years thanks to a Markov model.

The total duration of the study is 24 months (6 months of enrolment and 18 months of follow-up).

ELIGIBILITY:
Inclusion Criteria:

1. Adults with an atypical Hemolytic and Uremic Syndrome defined by at least 2 of the following parameters:

   * Thrombopenia (platelet count < 150 G/L)
   * Mechanical lytic anemia (Hb < 10 g/L, Lactate dehydrogenase > upper limit of normal, undetectable haptoglobin, presence of schistocytes on blood smear)
   * Acute renal failure
2. Eculizumab treatment

   * Without project of withdrawal in the next 18 months
   * Started since at least 6 months
   * Administrated with an unchanged administration schedule since at least 3 months (initial episode or relapse)
3. Atypical Hemolytic and Uremic Syndrome in remission
4. Patients who give informed consent.

Exclusion Criteria:

1. Patients on dialysis.
2. Women treated starting or planning a pregnancy.
3. Patients suffering from a typical or secondary microangiopathic hemolytic anemia (drugs, malignancies, autoimmune disease...)
4. Patients under protection of a judicial authority

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-10-20 (Actual); Primary Completion 2022-06-16 (Actual); Study Completion 2023-12-28 (Actual)

PRIMARY OUTCOMES:
Incremental Cost-Utility Ratio (ICUR) at 18 months of a personalized spacing of eculizumab infusions compared to the usual administration scheme without personalization, from the French health insurance perspective. | 18 months
  The ICUR will express the incremental cost per QALY (Quality-adjusted Life Years) gained over a 18-month time horizon. QALYs will be estimated from patient responses to the EQ-5D-5L instrument (EuroQol group - 5 Dimensions - 5 levels). Costs related to hospital care resources (medicalized information system program), transports (patient diary), eculizumab concentration dosing (cost estimation) will be estimated from the French Health Insurance perspective. Cost and QALY estimates will be used to estimate the within-trial ICUR.

SECONDARY OUTCOMES:
Incremental Cost-Utility Ratio at 5 years (incremental cost per QALY gained) of a personalized spacing of the eculizumab infusions compared to the usual administration scheme without personalization, estimated from a Markov model. | 5 years
  A Markov model will represent the patient's clinical progression across different health states over a 5-year period. Markov modelling will use the within-trial data to estimate the transition probabilities, the state cost and utility values.
Financial impact per year and over a 5-year period of a personalized spacing of eculizumab infusions | per year and over a 5-year period
  The financial impact of spreading the strategy of personalized spacing of eculizumab infusions, in patients in remission with atypical hemolytic uraemic syndrome requiring long-term treatment, will be estimated per year and over a 5-year period, from the French Health Insurance (using a budget impact model).
Quality of life measured over a 18-month period using different specific scales (KDQoL-SF, ReTransQoL-Version 2) dedicated to patients with renal disease | at baseline, 3, 6, 9, 12, 15 and 18 months.
  KDQoL-SF (Kidney Disease and Quality of Life™ Short Form) survey is a kidney-disease-specific quality of life instrument that assesses four domains : health, kidney disease, effects of kidney disease on daily life, satisfaction with care. Scores for each dimension are reported within the range 0-100, higher scores indicating better health- related quality of life.
  RTQ-V2 (ReTransQoL-Version 2) survey is a specific quality of life instrument for renal transplant recipients. It comprises of 32 items describing five domains: Physical Health, Social Functioning, Medical Care, Treatment and Fear of Losing Graft. Scores for each dimension are reported within the range 0-100, higher scores indicating better health- related quality of life.
  KDQoL-SF survey will be used for all patients, and RTQ-V2 survey for kidney transplant patients only. The quality of life will be measured every three months.
Determining the factors of intra- and inter- individual variability of eculizumab concentrations. | 5 years
  A study will be performed to determine whether biological and genetic (complement genetic variants reported as cause of HUS) parameters influence trough concentrations of eculizumab

CONTACTS AND LOCATIONS:
Locations (18):
- France (18):
  - CHU Amiens Picardie, Amiens
  - CHU d'Angers, Angers
  - Hôpital Tenon, APHP Tenon
  - CHU Besançon, Besançon
  - Hôpital de la Côte de Nacre, Caen
  - Hôpital Louis Pasteur, Chartres
  - Hôpital Gabriel Montpied, Clermont-Ferrand
  - Hospices Civils de Lyon, Lyon
  - Hopital de la conception, Marseille
  - Hôpitaux de Brabois, Nancy
  - Hotel Dieu, Nantes
  - Hopital Necker, Necker
  - Hopital Pasteur 2, Nice
  - Hôpital de la Milétrie, Poitiers
  - Hôpital Maison Blanche, Reims
  - Hôpital Pontchaillou, Rennes
  - Hôpital de Bois-Guillaume, Rouen
  - Nouvel Hôpital Civil, Strasbourg